CLINICAL TRIAL: NCT03683745
Title: Prevalence Survey for Innovative and Intensified Disease Management (IDM) Neglected Tropical Diseases (NTDs): A Cluster Randomised Two-stage Active Case Search for IDM-NTDs in Liberia
Brief Title: Integrated Mapping of Skin-presenting Neglected Tropical Diseases in Liberia
Status: Completed | Type: Observational
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: AIM Initiative (Unknown); Ministry of Health, Liberia (Other)
Responsible Party: Principal Investigator, Rachel Pullan, Associate Professor, London School of Hygiene and Tropical Medicine
Other Study IDs: 14698-1
Record Dates: First submitted 2018-09-19; First posted 2018-09-25 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Leprosy; Buruli Ulcer; Yaws; Lymphatic Filariases
Keywords: disease burden
MeSH Terms: conditions — Leprosy; Buruli Ulcer; Yaws; Elephantiasis, Filarial

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Specimens will be obtained from all clinically suspected cases, for confirmatory diagnosis. These include:
  * skin swabs of suspected yaws lesions
  * nasal swabs of suspected leprosy cases
  * skin swabs of Buruli ulcer lesions
  Samples will be tested using molecular analysis including PCR and sequencing for detection of T. pallidum, M. Ulcerans, M. leprae and other pathogens which can cause similar manifestations.
  Samples are to be stored (in Liberia, and in London) at -20 degrees in appropriately secured laboratory freezers (CL2 and CL3) for future research projects. This is explained in the information sheet, with a statement included in the consent forms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maryland: Maryland is a county in southeast Liberia. Survey clusters based on catchment populations served by community health volunteers (CHVs) around 24 district health facilities (primary sampling unit). Clusters will constitute ~600 people (~100 households) with population-weighted cluster selection applied. In total, 80 clusters will be required. CHVs would conduct house-to-house visits to develop a full census and listing of all possible cases using broad case definitions. Full details of all potential cases will then be passed to an expert verification team based at the closest health facility. Suspected cases will arrive at the health facility over a 10-day verification period to receive a diagnosis using clinical examination and/or laboratory confirmation.

SUMMARY:
Appropriate targeting of interventions for neglected tropical diseases (NTDs) that require innovative and intensified disease management (IDM) requires accurate data on the distribution of these diseases within endemic countries. In most instances however, existing case register data generated through national health management information systems or during programmatic activities do not provide an accurate representation of the true burden of IDM NTDs. This study will pilot a cluster randomized screening and confirmation survey to estimate the burden of IDM NTDs characterised by skin conditions associated with long-term disfigurement and disability. These include: leprosy, Buruli ulcer, yaws and lymphoedema and hydrocele resulting from lymphatic filariasis. The survey is being conducted in one county in Liberia.

The protocol involves community-level screening by community health volunteers trained to use photo-based visual aids to recognise changes in the skin that broadly indicates patent infection. All suspected cases will be verified in their homes by local and national experts trained in the diagnosis of skin-presenting NTDs. The survey will generate accurate district-level prevalence estimates of leprosy, yaws, Buruli ulcer and lymphatic filariasis-associated lymphoedema and hydrocele and quantify the total costs and cost per case detected. In addition, results from this protocol will be compared with routinely collected case register data, to better understand how health system records reflect the true disease situation on the ground and quantify unmet need.

DETAILED DESCRIPTION:
Innovative and intensified disease management (IDM) includes a range of different interventions - ranging from medicine to surgery - to relieve the symptoms and consequences of a group of neglected tropical diseases (NTDs) for which effective tools are scarce or where the widespread use of existing tools is limited. The World Health Organisation (WHO) has developed a series of strategies to achieve the control, elimination and eventual eradication of these NTDs, comprising universal access to early diagnosis and prompt treatment, improving active surveillance, integrating passive surveillance into health-service provision, and accelerating efforts towards elimination and eradication by intensifying core interventions. Appropriate targeting of IDM interventions requires accurate epidemiological data on the distribution of these NTDs within endemic countries. In most instances however, existing case register data generated through national health management information systems or during programmatic activities do not provide an accurate representation of the true burden of IDM NTDs.

A number of IDM NTDs are characterised by cutaneous manifestations that are associated with long-term disfigurement and disability. These include Buruli ulcer, cutaneous leishmaniasis, leprosy, mycetoma, yaws, onchocerciasis and lymphoedema and hydrocele (resulting from lymphatic filariasis and podoconiosis). These diseases require similar case-detection approaches, presenting opportunities for the development of novel, integrated mapping approaches. Population-based prevalence surveys (PBPS) are the gold standard methodology for obtaining accurate disease estimates when case detection and reporting through the health system is incomplete, and these have been used to provide sub-national estimates of disease distributions for yaws and podoconiosis. For less common outcomes (fewer than 1 case in 1000 individuals) however, standard PBPS rapidly become unfeasible. Given that the expected prevalence range for many of these IDM NTDs in endemic regions lies between as low as 1 in 10,000 for Buruli ulcer and 1-5% for yaws, it is clear that the PBPS approach requires adaptation to achieve the samples sizes needed to generate sufficiently precise prevalence estimates.

One alternative to randomly sampling individuals or households is to screen all residents within sampling clusters. House-to-house screening by mobile expert teams would likely yield the highest number of cases, but such a strategy would be expensive and difficult to sustain. As an alternative, trained village volunteers have been used during programmatic activities to effectively detect and refer diseases such as Buruli ulcer and leprosy in a number of countries. Given how difficult it is to diagnose many IDM-NTDs accurately, using community volunteers to perform an exhaustive house-to-house case search would require follow up expert case validation. The success of such an approach would thus rely on high levels of community awareness, coupled with well-trained village volunteers being able to recognise possible conditions, and a highly skilled, mobile case-validation team to confirm all potential cases. Effectively incorporating skill development in IDM-NTD screening among village volunteers could however represent a long-term and sustainable solution to the complex issue of managing these conditions at the community and primary health care level.

This study aims to establish the prevalence and distribution of case-management NTDs in the county of Maryland, Liberia using an integrated two-stage cluster-randomised sampling approach, including assessment of the proportion of cases not currently known to the health system.

The specific objectives include:

1. To generate regional prevalence estimates of (i) lymphatic filariasis-associated lymphoedema and hydrocele, (ii) yaws, (iii) Buruli ulcer and (iv) leprosy in Maryland, Liberia, including the proportion of cases not currently known to the health system
2. To model the endemicity status of (i) lymphoedema and hydrocele, (ii) yaws, (iii) Buruli ulcer and (iv) leprosy to support the development of targeted, integrated control strategies.
3. To compare case detection rates from active community-based screening and validation with passive case detection reported through routine health system reports and health management information systems.

This protocol represents a novel tool for integrated mapping of IDM-NTDs. These conditions are difficult to diagnose and lack effective tools for both case finding and disease management purposes. This strategy may provide a template for cost-effective case identification and management that can be integrated within routine health systems in similar epidemiological settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 must be willing and able to give informed consent for examination, and children over 13 years must be willing and able to give informed assent
* An adult (>18 year of age) parent or guardian must be present at the time of the examination who can give informed consent for children <18 years to be examined.

Exclusion Criteria:

* Individuals for whom no adult parent/guardian is available to provide consent and/or who are unwilling to provide assent/consent for themselves.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals resident in the study clusters, which were selected with probability proportional to size.
Sampling Method: Probability Sample
Enrollment: 56285 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Population prevalence of Lymphatic Filariasis | Over a four month period
  Clinical signs of lymphoedema and hydrocele associated with lymphatic filariasis
Population prevalence of Yaws | Over a four month period
  Clinical signs and PCR-confirmed yaws
Population prevalence of Buruli Ulcer | Over a four month period
  Clinical signs and PCR-confirmed Buruli ulcer

SECONDARY OUTCOMES:
Population prevalence of leprosy | Over a four month period
  Clinical signs of disease and of Grade 2 disability for leprosy
Population prevalence of BU and yaws in children | Over a four month period
  Clinical signs of Buruli ulcer and yaws in children <15years
Population prevalence of category 3 Buruli Ulcer | Over a four month period
  Category 3 lesions for Buruli ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Pullan, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Karsor Kollie, MSc, Principal Investigator — Ministry of Health, Liberia
Locations (1):
- Maryland County, Harper, Maryland County, Liberia

IPD SHARING:
Plan to Share IPD: Undecided